CLINICAL TRIAL: NCT01085032
Title: Transdermal Nicotine Therapy as an Adjunct to Behavioral Smoking Cessation Counseling in Syrian Primary Care Settings
Brief Title: Nicotine Patch Trial in Syrian Primary Care Settings
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Memphis (Other)
Responsible Party: Kenneth D. Ward, PhD, University of Memphis
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1R01DA024876 (NIH)
Record Dates: First submitted 2010-03-10; First posted 2010-03-11 (Estimated); Last update posted 2010-03-11 (Estimated); Status verified 2010-02

CONDITIONS: Smoking Cessation
Keywords: Smoking Cessation; Substance Withdrawal Syndrome; Depression
MeSH Terms: conditions — Smoking Cessation; Substance Withdrawal Syndrome; Depression | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): Behavioral Counseling and Nicotine Patch
  Interventions: Drug: Transdermal Nicotine
- Arm B (Placebo Comparator): Behavioral counseling and placebo patch
  Interventions: Drug: Placebo nicotine patch

INTERVENTIONS:
Drug: Transdermal Nicotine — Subjects in the experimental group receive six weeks of nicotine patch treatment, 24 hour dose, using a step-down algorithm. Participants who smoke greater than 10 cigarettes/day receive two weeks of 21 mg patch, followed by two weeks of 14 mg patch, and then two weeks of 7 mg patch. Participants who smoke 5-9 cigarettes per day receive four weeks of 14 mg patch, followed by two weeks of 7 mg.
  Arms: Arm A
Drug: Placebo nicotine patch — Subjects in the placebo condition receive an inert placebo patch matched for size, shape, color, and packaging.
  The same step-down dosing algorithm as in the experimental condition is used.
  Arms: Arm B

SUMMARY:
The study is a two-arm, parallel group, randomized, placebo-controlled, double blind trial, conducted at four primary health care centers in Aleppo, Syria, to test the efficacy of transdermal nicotine patch therapy vs. placebo patch therapy, when delivered with behavioral counseling, on smoking cessation rates.

DETAILED DESCRIPTION:
The study is a two-arm, parallel group, randomized, placebo-controlled, double blind trial, conducted at four primary health care centers in Aleppo, Syria, to test the efficacy of behavioral counseling with and without transdermal nicotine therapy on long-term smoking cessation rates. The trial will be conducted at four primary care clinics in Aleppo, Syria that are sponsored by private or non governmental organizations. Clinic physicians will be trained to provide a brief assessment of each patient's smoking status and motivation to quit, and to refer appropriate patients to a cessation clinic within the primary care center. Eligible and interested smokers will be randomized to receive behavioral cessation counseling + nicotine patch or behavioral cessation counseling + placebo patch. Behavioral counseling will be delivered by a physician at each clinic.

After eligibility is determined and a description of the cessation program has been provided, written informed consent will be obtained. When literacy is a concern, the consent form will be read to the subjects who will then mark the form to indicate consent.

Participants will provide baseline demographic data (age, gender, ethnicity, residence, marital status, education, occupation, income), smoking related information (smoking history, level of dependence, interest in quitting, comorbidities), and complete additional questionnaires to assess quitting self-efficacy, stage of change, withdrawal symptoms, and depression/mood.

Participants will then be allocated to one of two treatment conditions (Arm A: behavioral counseling + nicotine patch vs. Arm B: behavioral counseling + placebo patch) using random permuted blocks, stratified according to primary care center and gender. Specific behavioral and pharmacological intervention procedures are as follows:

Participants in Arm A will receive active transdermal nicotine, and participants in Arm B will receive placebo patch. Transdermal nicotine replacement was selected as the pharmacologic agent of choice, based on its ease of use, acceptability to patients, favorable side effect and contraindications profile, and its well researched and documented efficacy (Fiore et al., 1994). Additionally, our pilot intervention work in Syria indicates a high degree of acceptability of the patch as a potential smoking cessation intervention (Asfar et al., 2005).

In accordance with clinical practice guidelines in the U.S. (Fiore et al., 2000), participants will receive six weeks of patch treatment, 24 hour dose, using a step-down algorithm. Participants who smoke greater than 10 cigarettes/day will be receive two weeks of 21 mg patch, followed by two weeks of 14 mg patch, and then two weeks of 7 mg patch. Participants who smoke 5-9 cigarettes per day will receive four weeks of 14 mg patch, followed by two weeks of 7 mg.

Subjects in both arms receive three brief face-to-face counseling sessions and five brief (approximately 10 minute) phone counseling calls. Session 1 occurs 3-4 days before the scheduled quit day and focuses on preparing to quit. Calls 1 and 2 occur the day before and the day after quit day, respectively, and focus on surviving the first few days as a non-smoker. Session 2 takes place 7 days after the quit day and emphasizes provision of social support, problem solving, and coping with withdrawal symptoms and negative emotions. The final session occurs 14 days after quit day and emphasizes relapse prevention and coping skills training. An additional three phone calls occur 10, 30, and 45 days after quit day and provide social support, check progress, and reinforce coping skills. Follow-up assessments occur at 7 weeks, 6 months, and 12 months post-cessation.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* smoking continuously for at least one year and smoking 5 cigarettes every day
* Reside in the catchment area of one of the four primary care centers

Exclusion Criteria:

* diagnosed with a generalized dermatology disease, liver failure, hyperthyroidism, or pheochromocytoma
* current use of psychotropic drugs
* past year history of drug or alcohol abuse, unstable cardiovascular, psychiatric, or debilitating diseases based on physician assessment.
* currently pregnant, lactating, or intending to become pregnant in next 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2006-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Prolonged Abstinence | 7 weeks, 6 months and 12 months
  Self report and verified by exhaled CO levels of less than 10ppm. Prolonged abstinence will be defined as abstinence sustained after a 2 week grace period.

SECONDARY OUTCOMES:
7 day point prevalent abstinence | 7 weeks, 6 months and 12 months
  defined as non-smoking during the last 7 days and exhaled CO levels of <10ppm
Withdrawal symptoms | 7 weeks, 6 months, 12 months
  Measured with the Withdrawal Symptoms List (Hughes et al., 1986, 1991).
Depressive symptomatology | 7 weeks, 6 months, 12 months
  CES-D; Radloff, 1977

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth D Ward, PhD, Principal Investigator — University of Memphis
Locations (1):
- Four privately- or NGO-sponsored adult primary care clinics, Aleppo, Syria

REFERENCES:
- [Derived] Ward KD, Asfar T, Al Ali R, Rastam S, Weg MW, Eissenberg T, Maziak W. Randomized trial of the effectiveness of combined behavioral/pharmacological smoking cessation treatment in Syrian primary care clinics. Addiction. 2013 Feb;108(2):394-403. doi: 10.1111/j.1360-0443.2012.04048.x. Epub 2012 Nov 19. PMID 22882805